CLINICAL TRIAL: NCT03967314
Title: A Comparison of Ultrasound-Guided Modified-Thoracolumbar Interfacial Plane Block and Wound Infiltration for Postoperative Pain Management in Lumbar Spinal Surgery Patients
Brief Title: An mTLIP Block for Analgesia Management After Lumbar Spinal Surgery.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medipol University (Other)
Responsible Party: Principal Investigator, Bahadir Ciftci, Primary researcher, Medipol University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Medipol Hospital
Record Dates: First submitted 2019-05-22; First posted 2019-05-30 (Actual); Last update posted 2019-05-30 (Actual); Status verified 2019-05

CONDITIONS: Lumbar Disc Herniation
Keywords: Lumbar spinal surgery; Postoperative pain management; Modified thoracolumbar interfacial plane block
MeSH Terms: conditions — Intervertebral Disc Displacement | interventions — Sensitivity Training Groups

STUDY DESIGN:
Intervention Model Description: The patients were aged 18-65 years, American Society of Anesthesiologists classification I-II, and scheduled for lumbar disc surgery under general anesthesia. The patients were randomly divided into two groups using a randomizing computer program: a TLIP block group (group T) and a wound infiltration group (group W), with 30 patients in each group).
Who Masked: Participant, Outcomes Assessor
Masking Description: Outcomes Assessor and participant were blinded to the study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group T = TLIP block group (Active Comparator): After the induction of anesthesia and placement of the patient in a prone position, US-guided mTLIP block was performed via the lateral approach in group T. For postoperative analgesia, a dose of 1 g of paracetamol (IV) was administered routinely, every 8 h. All the patients received fentanyl via a patient-controlled analgesia device. The protocol was a 20 mcg bolus without an infusion dose, 20-min lockout time, and 4-h limit
  Interventions: Other: TLIP block group (group T)
- Group W = Wound infiltration group (Active Comparator): After the induction of anesthesia and placement of the patient in a prone position wound infiltration was performed in group W. For postoperative analgesia, a dose of 1 g of paracetamol (IV) was administered routinely, every 8 h. All the patients received fentanyl via a patient-controlled analgesia device. The protocol was a 20 mcg bolus without an infusion dose, 20-min lockout time, and 4-h limit
  Interventions: Other: Wound infiltration group (group W)

INTERVENTIONS:
Other: TLIP block group (group T) — In group T, the block was performed bilaterally under aseptic conditions using the US device with a high-frequency 12-MHz linear US probe. The probe was covered with a sterile sheath and placed vertically at the L3 vertebrae level. After visualizing the hyperechoic shadow of the spinous process and interspinous muscles as an anatomical guide point, the probe was moved forward in a lateral direction to visualize the longissimus and iliocostal muscles. Using the in-plane technique, a 22-G, 50-mm block needle was inserted between the muscles in a medial-to-lateral direction in the interfascial plane. Once the needle tip was placed within the interfacial plane and after careful aspiration to rule out intravascular needle placement, 2 ml of saline was injected to confirm the accuracy of the injection site. A dose of 0.25% bupivacaine (20 ml) was then injected in each side (total 40 ml).
  Arms: Group T = TLIP block group
Other: Wound infiltration group (group W) — In group W, a dose of 0.5% bupivacaine (20 ml) was injected for wound infiltration into the surgery site.
  Arms: Group W = Wound infiltration group

SUMMARY:
Pain management is an important issue following lumbar spinal surgery. Wound infiltration is a technique that a local anesthetic solution is infiltrated into the tissues around the surgical area. Modified thoracolumbar interfacial plane (mTLIP) block was described by Ahiskalioglu et al. In this study, the investigators aimed to compare the analgesic efficacy of the US-guided mTLIP block and wound infiltration following lumbar disc surgery.

DETAILED DESCRIPTION:
Spinal surgery in the lumbar region is one of the most common surgeries performed for leg and back pain. Postlumbar surgery pain can be severe and may progress to chronic pain during the postoperative period. Therefore, pain management is important after lumbar spinal surgery. Effective postoperative pain management enables early mobilization and shorter durations of hospital stays and may also reduce hospitalization-related complications, such as infections and thromboembolism.

There are a variety of techniques for postoperative pain management. These include intravenous-intramuscular injections, patient-controlled analgesia devices, local anesthetic infiltration, and regional anesthesia. Among these techniques, intramuscular and intravenous (IV) injections may be ineffective in pain management, as they are generally administered after the pain has commenced. In addition, intermittent treatment with analgesic agents may not result in a therapeutic level in the blood.

The most common analgesic agents used postoperatively are opioids. However, parenteral opioids may result in undesirable adverse events, such as nausea, vomiting, itching, sedation, and respiratory depression. Various methods are available to reduce the use of systemic opioids in postoperative pain management, one of which is local anesthetic infiltration (wound infiltration) into the operation site. Several studies reported that wound infiltration can reduce opioid consumption following surgery. Various regional anesthesia techniques can also be used to manage postoperative pain. Such techniques have a high success rate, especially if they are applied with ultrasound (US) guidance, as US improves visualization, thereby reducing potential complications. Previous research reported that US-guided modified thoracolumbar interfacial plane (mTLIP) block after lumbar spinal surgery via a lateral approach provided effective analgesia. No studies seem to have compared the analgesic effectiveness of wound infiltration versus TLIP block. In this study, the investigators compared the analgesic efficacy of the US-guided mTLIP block and wound infiltration following lumbar disc surgery. The primary aim was to compare postoperative opioid consumption. The secondary aim was to evaluate postoperative pain scores and adverse effects of opioids, such as allergic reactions, nausea, and vomiting.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) classification I-II
* Scheduled for lumbar discectomy/hemilaminectomy surgery under general anesthesia

Exclusion Criteria:

* Bleeding diathesis
* Receiving anticoagulant treatment
* Known local anesthetics and opioid allergy
* Infection of the skin at the site of the needle puncture
* Pregnancy or lactation
* Patients who do not accept the procedure

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2019-04-30 (Actual); Study Completion 2019-04-30 (Actual)

PRIMARY OUTCOMES:
Opioid consumption by the patients at postoperative 24 hours period | Postoperative 24 hours
  Fentanyl using

SECONDARY OUTCOMES:
Postoperative pain scores | Postoperative 24 hours period
  Postoperative pain assessment will be performed using the VAS score (0 = no pain, 10 = the most severe pain felt). The VAS scores at rest and during cough will be recorded at postoperative 0, 2, 4, 8, 16 and 24 hours.

CONTACTS AND LOCATIONS:
Overall Officials: Bahadir Ciftci, Asist.Prof, Principal Investigator — Medipol University
Locations (1):
- Istanbul Medipol University Hospital, Istanbul, Bagcilar, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared

REFERENCES:
- [Background] Ahiskalioglu A, Yayik AM, Alici HA. Ultrasound-guided lateral thoracolumbar interfascial plane (TLIP) block: Description of new modified technique. J Clin Anesth. 2017 Aug;40:62. doi: 10.1016/j.jclinane.2017.04.015. No abstract available. PMID 28625449
- [Background] Ahiskalioglu A, Alici HA, Selvitopi K, Yayik AM. Ultrasonography-guided modified thoracolumbar interfascial plane block: a new approach. Can J Anaesth. 2017 Jul;64(7):775-776. doi: 10.1007/s12630-017-0851-y. Epub 2017 Feb 27. No abstract available. PMID 28243853
- [Background] Gurbet A, Bekar A, Bilgin H, Korfali G, Yilmazlar S, Tercan M. Pre-emptive infiltration of levobupivacaine is superior to at-closure administration in lumbar laminectomy patients. Eur Spine J. 2008 Sep;17(9):1237-41. doi: 10.1007/s00586-008-0676-z. Epub 2008 Apr 19. PMID 18425538
- [Background] Kjaergaard M, Moiniche S, Olsen KS. Wound infiltration with local anesthetics for post-operative pain relief in lumbar spine surgery: a systematic review. Acta Anaesthesiol Scand. 2012 Mar;56(3):282-90. doi: 10.1111/j.1399-6576.2011.02629.x. Epub 2012 Jan 19. PMID 22260370